CLINICAL TRIAL: NCT02213601
Title: Efficacy of Yoga for Depressed Postpartum Women: A Randomized Controlled Trial
Brief Title: Efficacy of Yoga for Postpartum Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201105725
Record Dates: First submitted 2014-08-07; First posted 2014-08-11 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Depression, Postpartum
Keywords: Yoga; Complementary and Alternative Medicine Interventions; Treatment; Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum | interventions — Yoga

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yoga (Experimental): 8-week Gentle Vinyasa Flow yoga intervention
  Interventions: Behavioral: Yoga
- Wait-list Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Yoga
  Arms: Yoga

SUMMARY:
The aim of this project is to compare the efficacy of an 8-week yoga intervention, relative to a wait-list control (WLC) condition, for improving psychological functioning and health-related quality of life in depressed postpartum women. It was hypothesized that the yoga intervention would be significantly more efficacious than the wait-list control condition in reducing symptoms of depression and anxiety, and improving health-related quality of life, at the end of the 8-week yoga intervention.

ELIGIBILITY:
Inclusion Criteria:

* Score of 12 or greater on the 17-item Hamilton Depressing Rating Scale
* Participant must reside within a 30 mile radius of the yoga studios
* ≥ 6 weeks postpartum if delivery was either complicated and/or involved a cesarean section

Exclusion Criteria:

* Current or past diagnosis of bipolar disorder, schizophrenia or other psychotic disorder, alcohol or drug abuse/dependence (except nicotine), or anorexia in the past year
* Acute suicidal or homicidal risk
* Current mental health treatment, including psychotropic medications or psychotherapy with a certified therapist
* St. John's Wort or Fish oil
* Practiced yoga at a studio with a certified yoga instructor within the past month
* Significant medical disorder (e.g., seizure disorder) that is contraindicated for exercise in postpartum women

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2011-06; Primary Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in depression on the 17-item Hamilton Depression Rating Scale (HDRS) at week 8 | Baseline, Week 8
  The Hamilton Depression Rating Scale (HDRS) is a validated and reliable measure of the severity of depressive symptoms, and is used extensively in depression treatment studies. The 17-item HDRS is sensitive to treatment change in the postpartum population, and is a valid indicator of depression severity in postpartum depression despite the overlap between somatic HDRS items and typical experiences of postpartum women.

SECONDARY OUTCOMES:
Change from baseline in panic symptoms on the Inventory of Depression and Anxiety Symptoms Panic Scale (IDAS) at week 8 | Baseline, Week 8
  The Inventory of Depression and Anxiety Symptoms (IDAS) is a 64-item factor analytically derived, multidimensional inventory that uses a 5-point Likert scale to assess symptoms of depression and anxiety over the past 2 weeks (1 = not at all to 5 = extremely). The IDAS has strong internal consistency reliability, with median coefficient alphas greater than .80, and has been validated for use in a postpartum sample. The Panic scale is an 8-item measure that assesses symptoms traditionally linked to anxiety.
Change from baseline in social anxiety symptoms on the Inventory of Depression and Anxiety Symptoms Social Anxiety Scale (IDAS) at week 8 | Baseline, Week 8
  The Inventory of Depression and Anxiety Symptoms (IDAS) is a 64-item factor analytically derived, multidimensional inventory that uses a 5-point Likert scale to assess symptoms of depression and anxiety over the past 2 weeks (1 = not at all to 5 = extremely). The IDAS has strong internal consistency reliability, with median coefficient alphas greater than .80, and has been validated for use in a postpartum sample. The Social Anxiety scale is a 5-item measure that assesses symptoms traditionally linked to anxiety.
Change from baseline in traumatic intrusion symptoms on the Inventory of Depression and Anxiety Symptoms Traumatic Intrusions Scale (IDAS) at week 8 | Baseline, Week 8
  The Inventory of Depression and Anxiety Symptoms (IDAS) is a 64-item factor analytically derived, multidimensional inventory that uses a 5-point Likert scale to assess symptoms of depression and anxiety over the past 2 weeks (1 = not at all to 5 = extremely). The IDAS has strong internal consistency reliability, with median coefficient alphas greater than .80, and has been validated for use in a postpartum sample. The Traumatic Intrusions scale is a 4-item measure that assesses symptoms traditionally linked to anxiety.
Change from baseline in health-related quality of life symptoms on the Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) at week 8 | Baseline, Week 8
  The Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) is a well-validated measure of Health-related Quality of Life and consists of 36 items reflecting 8 domains of health: 1) role-limiting physical, 2) role-limiting emotional, 3) physical functioning, 4) social functioning, 5) mental health, 6) energy and vitality, 7) pain, and 8) general health perceptions.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa M Buttner, Ph.D., Principal Investigator — University of Iowa; Michael W O'Hara, Ph.D., Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

REFERENCES:
- [Background] Cooper PJ, Murray L, Wilson A, Romaniuk H. Controlled trial of the short- and long-term effect of psychological treatment of post-partum depression. I. Impact on maternal mood. Br J Psychiatry. 2003 May;182:412-9. PMID 12724244
- [Background] Da Costa D, Dritsa M, Rippen N, Lowensteyn I, Khalife S. Health-related quality of life in postpartum depressed women. Arch Womens Ment Health. 2006 Mar;9(2):95-102. doi: 10.1007/s00737-005-0108-6. Epub 2005 Oct 18. PMID 16231095
- [Background] Dennis CL. Influence of depressive symptomatology on maternal health service utilization and general health. Arch Womens Ment Health. 2004 Jul;7(3):183-91. doi: 10.1007/s00737-004-0053-9. Epub 2004 Jun 15. PMID 15241664
- [Background] Freeman MP. Complementary and alternative medicine for perinatal depression. J Affect Disord. 2009 Jan;112(1-3):1-10. doi: 10.1016/j.jad.2008.06.017. Epub 2008 Aug 8. PMID 18692251
- [Background] Gavin NI, Gaynes BN, Lohr KN, Meltzer-Brody S, Gartlehner G, Swinson T. Perinatal depression: a systematic review of prevalence and incidence. Obstet Gynecol. 2005 Nov;106(5 Pt 1):1071-83. doi: 10.1097/01.AOG.0000183597.31630.db. PMID 16260528
- [Background] Goodman JH. Women's attitudes, preferences, and perceived barriers to treatment for perinatal depression. Birth. 2009 Mar;36(1):60-9. doi: 10.1111/j.1523-536X.2008.00296.x. PMID 19278385
- [Background] O'Hara MW, Stuart S, Gorman LL, Wenzel A. Efficacy of interpersonal psychotherapy for postpartum depression. Arch Gen Psychiatry. 2000 Nov;57(11):1039-45. doi: 10.1001/archpsyc.57.11.1039. PMID 11074869
- [Background] Uebelacker LA, Epstein-Lubow G, Gaudiano BA, Tremont G, Battle CL, Miller IW. Hatha yoga for depression: critical review of the evidence for efficacy, plausible mechanisms of action, and directions for future research. J Psychiatr Pract. 2010 Jan;16(1):22-33. doi: 10.1097/01.pra.0000367775.88388.96. PMID 20098228
- [Background] Uebelacker LA, Tremont G, Epstein-Lubow G, Gaudiano BA, Gillette T, Kalibatseva Z, Miller IW. Open trial of Vinyasa yoga for persistently depressed individuals: evidence of feasibility and acceptability. Behav Modif. 2010 May;34(3):247-64. doi: 10.1177/0145445510368845. Epub 2010 Apr 16. PMID 20400694
- [Background] Wu P, Fuller C, Liu X, Lee HC, Fan B, Hoven CW, Mandell D, Wade C, Kronenberg F. Use of complementary and alternative medicine among women with depression: results of a national survey. Psychiatr Serv. 2007 Mar;58(3):349-56. doi: 10.1176/ps.2007.58.3.349. PMID 17325108
- [Background] Kinser PA, Bourguignon C, Whaley D, Hauenstein E, Taylor AG. Feasibility, acceptability, and effects of gentle Hatha yoga for women with major depression: findings from a randomized controlled mixed-methods study. Arch Psychiatr Nurs. 2013 Jun;27(3):137-47. doi: 10.1016/j.apnu.2013.01.003. Epub 2013 Apr 9. PMID 23706890
- [Background] Wisner KL, Perel JM, Peindl KS, Hanusa BH, Piontek CM, Findling RL. Prevention of postpartum depression: a pilot randomized clinical trial. Am J Psychiatry. 2004 Jul;161(7):1290-2. doi: 10.1176/appi.ajp.161.7.1290. PMID 15229064
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG; Consolidated Standards of Reporting Trials Group. CONSORT 2010 Explanation and Elaboration: Updated guidelines for reporting parallel group randomised trials. J Clin Epidemiol. 2010 Aug;63(8):e1-37. doi: 10.1016/j.jclinepi.2010.03.004. Epub 2010 Mar 25. PMID 20346624
- [Background] Ross LE, Gilbert Evans SE, Sellers EM, Romach MK. Measurement issues in postpartum depression part 1: anxiety as a feature of postpartum depression. Arch Womens Ment Health. 2003 Feb;6(1):51-7. doi: 10.1007/s00737-002-0155-1. PMID 12715264
- [Derived] Buttner MM, Brock RL, O'Hara MW, Stuart S. Efficacy of yoga for depressed postpartum women: A randomized controlled trial. Complement Ther Clin Pract. 2015 May;21(2):94-100. doi: 10.1016/j.ctcp.2015.03.003. Epub 2015 Apr 1. PMID 25886805